CLINICAL TRIAL: NCT06545136
Title: A Multicenter, Long-term, Follow-up Study to Investigate the Safety and Durability of Response Following Dosing of an Adeno-associated Viral Vector (FLT201) in Subjects With Gaucher Disease (GALILEO-2)
Brief Title: Long Term Follow-up Study of Type-1 Gaucher Subjects Post FLT201 Dose (GALILEO-2)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT201-02
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Gaucher Disease, Type 1
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dosed with FLT201 (Experimental)
  Interventions: Genetic: FLT201

INTERVENTIONS:
Genetic: FLT201 — FLT201 is a replication-incompetent single-stranded (ss) recombinant adeno-associated virus (AAV) vector. The vector is composed of a ss DNA genome packaged in an AAV-derived protein capsid.

SUMMARY:
This is a multicenter, long-term, follow-up trial of participants with Gaucher disease type 1 who received FLT201 treatment in a preceding clinical trial. Participants will be followed for 5 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants who have previously received FLT201 (including those who may have required recommencement or initiation of ERT/substrate reduction therapy [SRT]).
* 2. Participants able to give full informed consent and able to comply with all requirements of the trial.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) (including DLTs) | Week 38 to Month 60
  Treatment-emergent adverse events (including dose-limiting toxicities), with AEs graded per CTCAE version 5.0 (or later)

CONTACTS AND LOCATIONS:
Locations (4):
- Lysosomal Rare Disorders Research and Treatment Center, Fairfax, Virginia, United States
- Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre, Brazil
- Hospital Quironsalud Zaragoza, Zaragoza, Spain
- Salford Royal Hospital, Salford, United Kingdom